CLINICAL TRIAL: NCT01238731
Title: Persistence of Severe Pulmonary Artery Hypertension in Patients After vaLve replacemenT
Brief Title: Persistent Pulmonary Artery Hypertension After Valve Replacement
Acronym: SALT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: Actelion Pharmaceuticals Deutschland GmbH (Industry)
Responsible Party: Dr. Christoph Hammerstingl, Universitiy of Bonn, Medizinische Klinik und Poliklinik II
Other Study IDs: UKB_001_2010
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Persistent Severe PH After Valve Therapy
Keywords: Valve replacement; pulmonary hypertension; long term follow up
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Valve replacement: Patients undergoing valve replacement for severe valve disease will be screened for study entry

SUMMARY:
Background: Persistent severe pulmonary hypertension (PH) after mechanical valve replacement is a frequent finding in patients with severe valve-diseases. The reasons to develop PH are multifactorial and the prevalence of severe PH significantly worsens the patients´ outcome.

Aims: (i) To define the prevalence of PH in patients after valve replacement and (ii) to identify factors predicting persistent PH.

Methods: All patients which underwent valve replacement at our institution between the years 2008 -2010 will be screened retrospectively. Those patients with pre- procedural proven PH by means of right-heart catheterization will receive prospective follow-up with echocardiography. Diagnosis of persistent PH will be confirmed with right heart catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Proven pulmonary hypertension before valve replacement and informed consent for data acquisition

Exclusion Criteria:

* patients do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with proven PH before valve replacement by right heart catherterization will be screened for study entry.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-01 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Persistence of pulmonary hypertension after valve replacement for treatment of severe valve disease | > 6 months after valve therapy

SECONDARY OUTCOMES:
MACCE, all cause mortality during FU | Within 24 months after valve therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Klinik II, University of Bonn, Bonn, Germany